CLINICAL TRIAL: NCT04412941
Title: Myofascial Technique Combined With Myofunctional Exercises In Mild Obstructive Sleep Apnea-Hypopneas Syndrome: A Randomized Controlled Study
Brief Title: Respiratory Rehabilitation in Obstructive Sleep Apneas
Acronym: OSA20
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Collaborators: S. Spirito Hospital, Pescara, Italy (Unknown)
Responsible Party: Principal Investigator, Paolucci Teresa, Principal Investigator; Research fellow, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1837-28.06.2019
Record Dates: First submitted 2020-05-22; First posted 2020-06-02 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Sleep Disorder; Sleep Apnea Syndromes
Keywords: Rehabilitation; sleep obstructive apnea; oropharyngeal exercises; myofunctional exercises
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Myofunctional exercises + home oropharyngeal exercises + the rules of sleep hygiene
  Interventions: Behavioral: Myofunctional exercises; Behavioral: The rules of sleep hygiene
- Control group (Active Comparator): the rules of sleep hygiene
  Interventions: Behavioral: The rules of sleep hygiene

INTERVENTIONS:
Behavioral: Myofunctional exercises — Myofunctional exercises: Respiratory rehabilitation exercises with diaphragmatic breathing, thoracic mobilization exercises and manual pompage techniques, followed by manual trigger point therapy techniques, that were identified by palpation following the guidelines provided by Travell and Simons trigger point manual, the accessory inspiratory muscles like pectoralis minor muscle, scapula elevator muscle, Sternocleidomastoid muscle.
  Home oropharyngeal exercises: at every patient will be taught oropharyngeal exercises to perform at home twice a day (the duration of 15 minutes each session) involving in particular exercises for soft palate, tongue, facial and genio-glosso muscle.
  The rules of sleep hygiene: a list of behaviours that physiologically promote a good night's sleep.
  Other Names: home oropharyngeal exercises; the rules of sleep hygiene
  Arms: Treatment group
Behavioral: The rules of sleep hygiene — The rules of sleep hygiene: a list of behaviours that physiologically promote a good night's sleep.

SUMMARY:
The Obstructive Sleep Apnea is characterized by obstruction of the upper airway during sleep (for at least 10 sec), with repeated breathing pauses, accompanied by oxygen desaturation in the blood and by sleep interruption with repeated arousals.

The investigators hypothesized that good sleep hygiene, the execution of respiratory rehabilitation exercises, with specific myofascial exercises on the muscles that are compromised in the Obstructive Sleep Apnea, can improve the patient's clinical outcome and quality of life.

The objective of this study is to evaluate the effect of respiratory rehabilitation with myo-functional exercises in mild obstructive sleep.

DETAILED DESCRIPTION:
Patients: Eligible patients aged between 40 and 80 years old, with BMI < 30 and with a recent diagnosis of mild Obstructive Sleep Apnea evaluated with home night cardio-respiratory monitoring.

The investigators will exclude patients with one or more of the following conditions: subjects who regularly use hypnoinductive drugs, with craniofacial malformations, who have suffered recent facial trauma, suffering from hypothyroidism, suffering from neuromuscular diseases, with recent strokes, severe obstructive nasal disease, systemic infectious diseases and neoplastic diseases.

Home night cardio-respiratory monitoring: all patients will be evaluated according to international guidelines (AAMS American Academy Sleep Medicine) with an instrument equipped with sensors for detection oral/nasal flow, snoring, chest/abdomen movements, pulse oximetry and heart rate.

Questionnaire: The investigators will employ questionnaires validated in Italy: Snoring frequency (derived from the Berlin questionnaire); subjective daytime sleepiness (Epworth questionnaire); quality of sleep (Pittsburgh sleep quality questionnaire).

Patients will be randomized into two groups randomly with a 1: 1 ratio: group 1 (treated group) or group 2 (control group) for a total of 20 patients per group (according to the sample size calculation reported in the protocol).

The treatment group will be subjected to an integrated rehabilitation protocol, composed of Respiratory rehabilitation exercises with diaphragmatic breathing, thoracic mobilization exercises and manual pompage techniques, followed by manual trigger point therapy techniques, (that were identified by palpation following the guidelines provided by Travell and Simons trigger point manual), the accessory inspiratory muscles like pectoralis minor muscle, scapula elevator muscle, Sternocleidomastoid muscle. The integrated rehabilitation protocol will be 45 minutes, 3 weekly sessions for 4 weeks, for a total of 12 consecutive sessions. Also, at every patient will be taught oropharyngeal exercises to perform at home twice a day (the duration of 15 minutes each session) involving in particular exercises for soft palate, tongue, facial and genio-glosso muscle.

Both in the treated group and the control group will be given a booklet with the rules for proper sleep hygiene because sleep is influenced by our lifestyle and various environmental factors can affect the quality of night sleep.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild Obstructive Sleep Apnea (5≤AHI≤14)
* age between 40 and 80 years
* BMI <30.

Exclusion Criteria:

* regular use of Hypno-inducing drugs,
* severe nasal obstructive disease,
* primary pulmonary pathology,
* craniofacial malformations,
* recent facial traumas,
* hypothyroidism,
* neuromuscular diseases,
* recent stroke,
* systemic infectious diseases,
* neoplastic diseases.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in apnea/hypopnea index (AHI) | 4 months
  AHI is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep.
Sleep questionnaires, Berlin Questionnaire | 4 months
  it consists of 3 categories related to the risk of sleep apnea (1-severity of snoring, 2- excessive daytime sleepiness, 3-history of obesity or high blood pressure). Depending on the answers and therefore the reported symptoms, it allows a subdivision in high risk or low risk of having apneas;
Sleep questionnaires, Epworth Sleepiness Scale | 4 months
  it is a scale intended to measure daytime sleepiness with a short questionnaire; the answers range from normal (0) to intense (3) in eight different situations; a total score greater than 10 is considered excessive daytime sleepiness
Sleep questionnaires, Pittsburgh Sleep Quality Index | 4 months
  It is a self-administered questionnaire that assesses sleep quality over a 1-month time interval. Evaluate seven sleep items on a scale of 0 to 3, 0 indicating no difficulty and 3 indicating severe difficulty. The results are expressed in an overall score (between 0 and 21). Values above 5 are consistent with poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Paolucci, MD, PhD, Principal Investigator — University G.d'annunzio - Chieti Pescara
Locations (1):
- Teresa Paolucci, Chieti, Abruzzo, Italy

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available, because we didn't get organized